CLINICAL TRIAL: NCT01118611
Title: A Cancer Research UK Phase I Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Aurora B Inhibitor GSK1070916A in Patients With Advanced Solid Tumors
Brief Title: Aurora B/C Kinase Inhibitor GSK1070916A in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000669923; CRUK-CR0802-11; EUDRACT-2008-005031-15
Record Dates: First submitted 2010-04-14; First posted 2010-05-06 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: Aurora B/C kinase inhibitor GSK1070916A
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: diffusion-weighted magnetic resonance imaging + PET CT
Radiation: fludeoxyglucose F 18 dynomic contrast

SUMMARY:
RATIONALE: Aurora B/C kinase inhibitor GSK1070916A (GSK1070916A) may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of GSK1070916A in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine and establish the safety profile of Aurora B/C kinase inhibitor GSK1070916A and define the dose-limiting toxicity in patients with advanced solid tumors.
* To determine the maximum-tolerated dose of Aurora B/C kinase inhibitor GSK1070916A in these patients.

Secondary

* To determine plasma pharmacokinetic (PK) parameters following administration of Aurora B/C kinase inhibitor GSK1070916A in these patients.
* To evaluate tumor response after at least 1 cycle of treatment with Aurora B/C kinase inhibitor GSK1070916A in these patients.
* To propose a safe dose for Phase II evaluation.

Tertiary

* To investigate the effects of Aurora B/C kinase inhibitor GSK1070916A on markers of mitosis/cell proliferation and apoptosis in humans.
* To investigate the metabolism of Aurora B/C kinase inhibitor GSK1070916A in humans.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive Aurora B/C kinase inhibitor GSK1070916A IV over 1 hour once daily on days 1-5. Courses repeat every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients receive escalating doses of Aurora B/C kinase inhibitor GSK1070916A until the maximum-tolerated dose (MTD) is determined. Once the MTD has been defined, 15-18 additional patients are recruited for an expanded MTD cohort in which patients receive Aurora B/C kinase inhibitor GSK1070916A at the MTD. Patients at the expanded MTD cohort must consent to have either tumor biopsies taken or FDG-PET/CT and DW-MRI scans performed.

Patients may undergo tissue, blood, and urine sample collection periodically for pharmacokinetic, pharmacodynamic, and other correlative laboratory studies.

After completion of study therapy, patients are followed up for 28 days.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
Eligibility criteria The patient must fulfil the eligibility criteria (listed in Section 4.1.1 and 4.1.2).

Additional eligibility criteria must be fulfilled for the expanded MTD cohort (listed in Section 4.1.3).

4.1.1 Inclusion criteria:

1. Histologically or cytologically proven solid tumour refractory to conventional treatment, or for which no conventional therapy exists
2. Life expectancy of at least 3 months
3. World Health Organisation (WHO) performance status of 0 or 1
4. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day -1) before the patient goes on study. Laboratory Test Value required Haemoglobin (Hb) ≥ 10.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) AND aspartate aminotransferase (AST) ≤ 2.5 x ULN unless raised due to tumour in which case up to 5 x ULN is permissible Calculated creatinine clearance (preferably measured by EDTA/ DTPA (isotope method) otherwise to be calculated using Wright formula) ≥ 50 mL/min (uncorrected value)
5. 18 years or over
6. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up

4.1.2 Exclusion criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C and six weeks for investigational medicinal products) before treatment.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the Drug Development Office (DDO) should not exclude the patient.
3. Known brain metastases.
4. Patients on therapeutic anti-coagulation with warfarin are excluded. (1mg warfarin for line maintenance is acceptable; conversion to low molecular weight heparin is acceptable but must be done a minimum of seven days prior to the first dose of study drug).
5. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have a intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
6. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (e.g. condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
7. Major thoracic or abdominal surgery from which the patient has not yet recovered.
8. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
9. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
10. QTc interval ≥ 450 msecs for men and ≥ 470 msecs for women or other clinically significant electrocardiogram (ECG) abnormalities (QTc preferably calculated using the algorithm in Appendix 6).
11. Use of medicines known to prolong QTc within 14 days prior to the first dose of study drug (see Category 1 of Appendix 5).
12. Previous exposure to aurora kinase inhibitors
13. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA] - refer to Appendix 4)
14. History of cardiac ischaemia, cardiac arrhythmias, coronary angioplasty or stenting in the previous 12 months. Patients currently on medication for cardiac arrhythmias are also excluded.
15. Patients with a known left ventricular ejection fraction (LVEF) <50%. A multi-gated acquisition (MUGA) scan or echocardiogram must be performed if clinically indicated.
16. Any other condition which in the Investigator"s opinion would not make the patient a good candidate for the clinical trial.
17. Is a participant or plans to participate in another interventional clinical study, whilst taking part in this Phase I study of GSK1070916A. Participation in an observational study would be acceptable.

4.1.3 Additional inclusion / exclusion criteria for expanded MTD cohort:

Once tolerability has been confirmed in the initial three to six patients of the MTD, further patients in this expanded cohort must either consent to have tumour biopsies taken or having FDG PET-CT and DW/DCE-MRI scans performed. The minimum number of patients required in each part of the expansion cohort is six. The following additional inclusion / exclusion criteria will apply.

For patients consenting to tumour biopsies:

1. Additional written (signed and dated) informed consent for tumour biopsies must be given.
2. The patient"s tumour should be amenable to biopsy.

   For patients consenting to FDG PET-CT and DW/DCE-MRI scans:
3. Additional written (signed and dated) informed consent for FDG PET-CT and DW/DCE-MRI scans must be given.
4. Patients with diabetes must have their condition under good control (blood sugar less than 10mmol/L).
5. Patients must be able to tolerate / comply with imaging protocol (i.e. patients with high levels of pain, urinary incontinence, or claustrophobia etc should be excluded).
6. Patients with tumours known to be poorly FDG avid (e.g. mucinous adenocarcinoma, well differentiated neuroendocrine or hepatocellular carcinoma) or falsely negative (e.g. all tumours less than 5-6mm) are excluded. Refer to Appendix 7 for full list of excluded tumours.
7. Patients with implanted metallic devices (e.g. pacemaker) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Causality of each adverse event to Aurora B/C kinase inhibitor GSK1070916A and grading severity according to NCI CTCAE Version 4.02
Maximum-tolerated dose (MTD)

SECONDARY OUTCOMES:
Measurement of PK parameter values for Aurora B/C kinase inhibitor GSK1070916A including AUC, Cmax, Tmax, and half life (all cohorts)
Response assessment (stable disease, partial response, or complete response)
Analysis of phosphohistone H3, Ki67, and cleaved caspase 3 in skin-punch biopsies (all cohorts) and tumor biopsies (at the MTD only)
Analysis of caspase-cleaved cytokeratin 18 in serum samples (all cohorts)
Investigation of metabolite concentration in samples of blood (all cohorts) and urine (at the MTD only)
Safe dose for phase II evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, BMedSci, FRCP, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital
Locations (2):
- United Kingdom (2):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Barts and the London School of Medicine, London, England